CLINICAL TRIAL: NCT00699439
Title: A Reminder System for Paper-Based Asthma Guidelines in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 070206
Record Dates: First submitted 2008-06-12; First posted 2008-06-18 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Asthma; Medical Informatics
Keywords: Medical Informatics; Asthma; Emergency Service, Hospital; Bayesian Method
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): If a patient is identified as having an asthma exacerbation by the Bayesian Network, the paper-based flow-chart will be printed out to place on the chart.
  Interventions: Other: Paper-based asthma flow diagram
- B (No Intervention): If a patient is identified as having an asthma exacerbation by the Bayesian Network, and assigned to the control group, no flow-chart will be printed out.

INTERVENTIONS:
Other: Paper-based asthma flow diagram — If a patient is identified as having an asthma exacerbation by the Bayesian Network, the patients will be randomized to either arm A or B. If in A, the paper-based flow-chart will be printed out to place on the chart.
  Arms: A

SUMMARY:
The primary idea is that the use of a computerized reminder system to help with the guideline implementation will increase utilization and adherence of guideline-driven care, leading to improved patient outcomes. The hypothesis we aim to address is that an automatic, computerized reminder system for detecting asthma patients in the pediatric ED will increase paper-based guideline utilization compared to paper-based guideline without the system.

We aim to implement a real-time, computerized asthma detection system and integrate the system with the pediatric emergency department information system, and evaluate the effect of the asthma detection system on reminding clinicians to use the paper-based asthma guideline.

DETAILED DESCRIPTION:
Asthma is the leading chronic childhood disease affecting 9 million children (12.5%) under 18 years of age (1). Asthma exacerbations cause an estimated 14 million missed school days (2) and more than 1.8 million emergency department (ED) visits annually (2), and account for >60% of asthma-related costs (3). The chronic characteristic of asthma carries a considerable economic burden.

Uncontrolled asthma can lead to exacerbations requiring the patient to seek immediate care, frequently in an ED setting. Several asthma guidelines, including the nationally accepted guideline from the National Heart, Lung, and Blood Institute (NHLBI), exist to support clinicians in providing adequate treatment. Utilization of and adherence with asthma guidelines improves patients' clinical care (4, 5). However, guideline adherence remains suboptimal. In the ED, early recognition and accurate assessment of the severity of airway obstruction and response to therapy are fundamental to the improvement of health for patients with asthma. The NHLBI guidelines emphasize early recognition and treatment of asthma exacerbations, as well as appropriate treatment stratified by severity.

Computer applications for patient care can address barriers to optimal medical care. Computer systems have improved the use and adherence to practice guidelines, provide clinical alerts and reminders, and generate patient-specific treatment recommendations and educational material. Implementation of guideline-driven decision support is frequently paper-based or computerized. In either form a major barrier remains on the busy clinicians to remember to initiate the guideline a process and to embed the guideline tasks in the clinical workflow of the care team (5). The proposed study examines the benefits of a novel approach for reminding clinicians in an ED setting to use guideline-driven care. The approach will apply a workflow-embedded process taking advantage of an advanced information technology infrastructure. The informatics approach will include two elements: a) a computerized, real-time reminder system, which will automatically detect guideline-eligible patients without requiring additional data entry, and b) a computerized, workflow-embedded guideline implementation.

References

1. Ref: QuickStats: Percentage of Children Aged <18 years Who Have Ever Had Asthma Diagnosed, by Age Group --- United States, 2003; MMWR April 29, 2005 / 54(16);412. http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5416a5.htm
2. Allergy & Asthma Advocate. Quarterly patient newsletter of the American Academy of Allergy, Asthma and immunology. 2004.
3. Grimshaw JM, Eccles MP, Walker AE, Thomas RE. Changing physicians' behavior: what works and thoughts on getting more things to work. J Contin Educ Health Prof. 2002;22:237-243.
4. National Heart, Lung, and Blood Institute, National Asthma Education and Prevention Program. Expert Panel Report 2: Guidelines for the diagnosis and management of asthma. 1997.
5. Scribano PV, Lerer T, Kennedy D, Cloutier MM. Provider adherence to a clinical practice guideline for acute asthma in a pediatric emergency department. Acad Emerg Med. 2001;8:1147-1152.

ELIGIBILITY:
Inclusion Criteria:

The study's inclusion criteria are:

* All patients aged 2-18 years;
* Emergency Severity Index 2 to 5; AND
* Availability of completed computerized triage documentation.

Exclusion Criteria:

The exclusion criteria are:

* Critically ill patients (Emergency Severity Index 1)
* Patients who leave-without-being seen
* Patients who leave against-medical-advice
* Patients whose final diagnosis was not asthma (false positive identification by the detection system) or were determined not to be eligible for the guideline.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1102 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Guideline utilization. Guideline utilization will be defined as having used the guideline for the documentation of at least one assessment (asthma score). | Within 1 week after visit
Guideline Adherence. The measurement of guideline adherence includes three measures: a) asthma assessment (score); b) treatment compatible with assessment (or documentation of reason to deviate); and c) adherence to guideline schedule. | Within 1 week after visit

CONTACTS AND LOCATIONS:
Overall Officials: Judith W Dexheimer, MS, Principal Investigator — Vanderbilt University; Dominik Aronsky, MD, PhD, Principal Investigator — Vanderbilt University; Donald H Arnold, MD, MPH, Study Chair — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Dexheimer JW, Brown LE, Leegon J, Aronsky D. Comparing decision support methodologies for identifying asthma exacerbations. Stud Health Technol Inform. 2007;129(Pt 2):880-4. PMID 17911842
- [Background] Sanders DL, Aronsky D. Prospective evaluation of a Bayesian Network for detecting asthma exacerbations in a Pediatric Emergency Department. AMIA Annu Symp Proc. 2006;2006:1085. PMID 17238704
- [Background] Sanders DL, Aronsky D. Detecting asthma exacerbations in a pediatric emergency department using a Bayesian network. AMIA Annu Symp Proc. 2006;2006:684-8. PMID 17238428
- [Background] Sanders DL, Gregg W, Aronsky D. Identifying asthma exacerbations in a pediatric emergency department: a feasibility study. Int J Med Inform. 2007 Jul;76(7):557-64. doi: 10.1016/j.ijmedinf.2006.03.003. Epub 2006 May 2. PMID 16647876